CLINICAL TRIAL: NCT03607123
Title: Stepwise Atrial Fibrillation supprEssion Treatment in Patients With Paroxysmal Atrial Fibrillation and Sinus Node Dysfunction: Intensive Device Follow-up
Brief Title: Atrial Fibrillation With Sinus Node Dysfunction: Intensive Device Follow-up
Acronym: SAFE PAF-SND
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Vice Director of Division of Cardiology, The First Affiliated Hospital of Nanjing Medical University; Professor of Medicine, Nanjing Medical University, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2017-SR-235.A2
Record Dates: First submitted 2018-07-08; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Sinus Node Dysfunction; Atrial Fibrillation
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Baseline: After implantation of pacemaker, the pacing mode and the lower rate of pacemaker will be set as VDD and 50/45 bpm respectively, to get the baseline burden of atrial fibrillation without atrial pacing. Except for beta-blockers digoxin, and CCB to control heart rate, anti-arrhythmic drugs (AAD) will not be prescribed. Patients who can not tolerate will drop out. After follow-up of at least 3 month, patients with AF lasting longer than one minute detected by pacemaker will go to next group / stage (Atrial Pacing, Step1).
  Interventions: Other: programing of pacemaker
- Atrial Pacing (Step 1): After Baseline and after follow-up of at least 3 month, patients with AF lasting longer than one minute detected by pacemaker will come to this group /stage (Atrial Pacing). At this stage, the pacing mode and the lower rate of pacemaker will be set as DDD and 70/60 bpm respectively, to perform relatively high-rate atrial pacing. Except for beta-blockers digoxin, and CCB to control heart rate, anti-arrhythmic drugs (AAD) will not be prescribed. After follow-up of at least 3 month, patients with AF lasting longer than one minute detected by pacemaker will go to next group/stage (AAD, Step1).
  Interventions: Other: programing of pacemaker
- AAD (Step 2): After Step 1, and after follow-up of at least 3 month, patients with AF lasting longer than one minute detected by pacemaker will come to this group/stage. Anti-arrhythmic drugs including propafenone, amiodarone and dronedarone will be prescribed. After follow-up of at least 6 month, patients with AF lasting longer than one minute detected by pacemaker will go to next group/stage (RFCA, Step3).
  Interventions: Procedure: AF ablation
- RFCA (Step 3): After Step 2, and after follow-up of at least 6 month, patients with AF lasting longer than one minute detected by pacemaker will come to this group/stage (RFCA, Step3). Patients will receive catheter ablation of AF, up to patients' willingness. After follow-up of at least 12 month, patients without AF lasting longer than one minute detected by pacemaker will go to next group/stage (SAFE PAF-SND II).
  Interventions: Procedure: AF ablation; Drug: Anti arryhthmic drugs
- SAFE PAF-SND II: After RFCA, and after follow-up of at least 12 month, patients without AF lasting longer than one minute detected by pacemaker will come to this group/stage (SAFE PAF-SND II). At this stage, the pacing mode and the lower rate of pacemaker will be set as VDD and 40 bpm respectively. If the patient can not tolerate, the the pacing mode and the lower rate of pacemaker will be set as DDD/DDDR and 60 bpm. If the patient has no symptom related to bradycardia, he/she will be followed up until the end of this study.
  Interventions: Other: programing of pacemaker; Procedure: AF ablation

INTERVENTIONS:
Other: programing of pacemaker — Different programing parameters will be set in different group/stage
  Groups: Atrial Pacing (Step 1); Baseline; SAFE PAF-SND II
Procedure: AF ablation — AF ablation can only be performed in Step 3
  Groups: AAD (Step 2); RFCA (Step 3); SAFE PAF-SND II
Drug: Anti arryhthmic drugs — Anti arryhthmic drugs can be prescribed in Step 2, Step3 and SAFE PAF-SND
  Groups: RFCA (Step 3)

SUMMARY:
The study will try to access the efficacy of atrial pacing, medication and radiofrequency ablation in treating patients with paroxysmal atrial fibrillation and sinus node dysfunction; to identify the response to these treatments in patients with "functional" and organic sinus node dysfunction respectively; to explore the necessity of pacemaker implantation in patients with "functional" sinus node dysfunction. Patients who meet the inclusion criteria will receive pacemaker implantation followed by trial pacing, medication and radiofrequency ablation of AF. Device data will be analyzed to answer the question. And after follow-up of 1 year, lower rate of pacemaker will be set as 40 bpm for patients without AF. The proportion of pacing and patients' tolerance will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 - 80 years
* Longest RR interval ≥ 3 seconds in sinus rhythm or when atrial arrhythmia (atrial fibrillation/atrial arrhythmia/atrial flutter) is converted to sinus rhythm (documented by either holter monitor or electrogram).
* Meet the indications of permanent pacemaker implantation in patients with SND according to the 2012 ACCF/AHA/HRS Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities.
* Evidence of paroxysmal atrial fibrillation ( two or more symptomatic episodes within 6 months)
* Willing to sigh informed consent

Exclusion Criteria:

* Type II second-degree or three-degree atrioventricular block (in sinus rhythm)
* Intrinsic PR interval ≥ 300 ms in sinus rhythm
* Persistent AF（including long-standing persistent AF）
* Severe structural heart disease(e.g. ischemic heart disease that requires revascularization, rheumatic heart disease that requires valve replacement, cardiomyopathy except hypertensive myocardial hypertrophy)
* Work high above the ground or heavy physical labour
* Malignant ventricular arrhythmias
* New York Heart Association (NYHA) class III or IV
* AF secondary to electrolyte imbalance, thyroid dysfunction, vasovagal reaction or other reversible or non-cardiac causes
* Previous procedures dealing with AF (including radiofrequency ablation and surgical operation)
* Cardiac implantable electronic device implantation history
* Severe hepatic and renal dysfunction(serum creatinine above the upper normal limit of the center, or chronic renal dysfunction ; ALT or AST more than 2 times the upper normal limit of the center, or bilirubin more than 2 times the upper normal limit of the center, or hepatic cirrhosis)
* Contraindication to propafenone/amiodarone/dronedarone(except bradycardia)
* Contraindication to oral anticoagulants
* Women who are pregnant
* Presence of malignant tumor
* Severe coagulation disorder (without any anticoagulation treatment)
* The investigators do not think the patient is eligible for this study
* Patient is unwilling to cooperate with the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the Eligibility Criteria will be enrolled. The anticipated number of patients is 200.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2022-07-04 (Estimated); Study Completion 2022-07-04 (Estimated)

PRIMARY OUTCOMES:
proportion of ventricular pacing | through study completion, an average of 2 years

SECONDARY OUTCOMES:
symptom related to bradycardia | through study completion, an average of 2 years
AF burden | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided